CLINICAL TRIAL: NCT03875209
Title: A Phase 1 Dose-escalation Study of the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of the Bispecific Antibody 10E8.4/iMab in HIV-1-infected and Uninfected Individuals
Brief Title: 10E8.4/iMab Bispecific Antibody in HIV-uninfected and HIV-infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Ho (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); International AIDS Vaccine Initiative (Network); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, David Ho, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAS1239
Record Dates: First submitted 2018-10-02; First posted 2019-03-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Intervention Model Description: Dose escalation, open-label (IV or SC administration), placebo-controlled (SC administration)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants in SC dosing Arm 4 Groups J and K will be blinded as will providers and members of the study site team. Study pharmacists will not be blinded. Safety monitoring committee will not be blinded. All participants treated IV and participants treated 1 mg/kg SC will not be masked (open-label).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: 10E8.4/iMab IV or SC HIV- (Experimental): Arm 1; Groups A-C; 3 dosing groups: HIV-uninfected individuals
  Interventions: Biological: 10E8.4/iMab
- Arm 2: 10E8.4/iMab IV HIV- (Experimental): Arm 2; Groups D-F; 3 dosing groups: HIV-uninfected individuals
  Interventions: Biological: 10E8.4/iMab
- Arm 3 and 3a: 10E8.4/iMab IV HIV+ (Experimental): Arm 3; Group H; 1 dosing group: HIV-infected individuals with HIV-1 RNA levels between 1,000 and 100,000 copies/mL and cluster of differentiation 4 (CD4)>350 cells/mm3; Arm 3a; Group I; 1 dosing group: HIV-infected and suppressed individuals
  Interventions: Biological: 10E8.4/iMab
- Arm 4: 10E8.4/iMab SC HIV- (Experimental): Arm 4; Groups J and K: HIV-uninfected individuals
  Interventions: Biological: 10E8.4/iMab

INTERVENTIONS:
Biological: 10E8.4/iMab — bispecific monoclonal antibody

SUMMARY:
Many HIV-infected individuals mount a broad neutralizing serologic response 2-3 years after infection. Broadly neutralizing antibodies might play an important role in protection from acquisition of HIV infection because they can protect macaques from infection, and the presence of anti-HIV antibodies was the only positive correlate of protection in an HIV vaccine efficacy trial (RV144 trial). HIV neutralizing antibodies also have the potential to alter the course of HIV infection in humans. Therefore, these antibodies might be useful to both prevent and treat HIV-1 infection.

This is a phase 1 dose escalating clinical trial to evaluate the safety, tolerability, pharmacokinetics and the antiretroviral effects of a novel bispecific monoclonal antibody 10E8.4/iMab in HIV-infected and HIV-uninfected individuals. The study will be conducted as a multi-center study at the Columbia University Medical Center in New York City and the Orlando Immunology Center in Orlando, Florida.

DETAILED DESCRIPTION:
There are 4 study Arms as it is possible that pharmacokinetics (PK) may differ between HIV-1-uninfected individuals (Arms 1, 2 and 4) and HIV-1-infected and viremic individuals (Arm 3). Safety and tolerability as well as PK may differ between the IV and SC routes, Arms 1, 2 and 4.

A dose escalation design has been used to establish safety and tolerability at very low doses of 10E8.4/iMab as this is a first in man study. Once demonstrated, dose levels would be increased to dosing levels thought to be more clinically relevant.

The numbers of subjects receiving active antibody in each study arm are relatively balanced such that an initial evaluation of the primary endpoint with additional dosing to provide insights into both PK and antiviral activity as well as some exploratory endpoints such as immunogenicity will be possible.

This study is a phase 1 clinical trial to evaluate the safety and tolerability, pharmacokinetics and the antiretroviral activity of the bispecific monoclonal antibody 10E8.4/iMab in HIV-infected and HIV-uninfected individuals.

HIV uninfected, healthy volunteers will be administered either one intravenous infusion of 10E8.4/iMab at one of five increasing dose levels (0.3 mg/kg, 1 mg/kg, 3 mg/kg, 10 mg/kg and 30 mg/kg) or one SC injection of 1 mg/kg, 2.5 mg/kg or 10 mg/kg or placebo and will be followed for 24 weeks after 10E8.4/iMab administration. HIV-infected volunteers will be administered one intravenous infusion of 10E8.4/iMab at one of three increasing dose levels (3 mg/kg, 10 mg/kg and 30 mg/kg).

Arm 1 consists of 3 groups: Group A: 0.3 mg/kg IV, N=3; Group B: 1mg/kg SC, N=3; and Group C: 1mg/kg IV, N=3. All HIV-1 uninfected, dosed once.

Arm 2 consists of 3 groups: Group D: 3mg/kg, N=6; Group E: 10mg/kg, N=6; and Group F: 30 mg/kg, N=6. All HIV-1 uninfected, dosed IV once.

Arm 3 consists of 2 groups: H: 10mg/kg, N=4 and Group I: 30 mg/kg, N=4. All HIV-1 infected, dosed IV once.

Arm 4 consists of 2 groups: Group J: 2.5 mg/kg, N=9, 6 active, 3 placebo; Group K: 10mg/kg, N=9, 6 active, 3 placebo, dosed SC once.

Since the safety and tolerability profiles, as well as the PK profile might differ between HIV-infected and HIV-uninfected individuals, dose-escalation is planned in both study populations. Dosing in Arm 1 Groups A, B and C; Arm 2 Groups D and E; and Arm 4 Groups J and K will be done prior to initiation of dosing in Arm 3 due to safety considerations.

Arm 3 will include HIV-infected individuals off antiretroviral therapy (ART) for at least 4 weeks with plasma HIV-1 RNA levels < 100,000 copies/ml (both ART naïve and individuals that discontinued ART due to intolerance or by choice can be included in this group), or HIV-infected individuals on stable ART with plasma HIV-1 RNA levels > 1000 copies/ml.

The stated numbers of participants are the minimal number per dosing group. A safety monitoring committee may request additional enrollment in a specific Arm or Group based on the occurrence of dose limiting toxicities defined as any Grade 3 or greater adverse event that is probably or definitely related to the investigational product.

Study visits are all outpatient and include:

1. a screening phase of up to 2 visits
2. an administration visit at which 10E8.4/iMab is given either IV or SC in doses based on body weight and specific Arm and Group assignment.
3. follow up visits that will occur at days 2, 7, 10 and weeks 2, 3, 4, 6, 8, 12 and 24. Subjects who received placebo SC may not be required to return for the week 24 visit.

ELIGIBILITY:
Inclusion Criteria for HIV uninfected volunteers: Arms 1, 2 and 4:

* Healthy volunteers born male and female as assessed by medical history and physical examination
* Aged >18 and <60 years at the time of screening
* Ability and willingness to provide written informed consent
* Willingness to comply with protocol schedule
* Willingness to undergo HIV-1 testing
* Non-reactive 4th generation point of care HIV-1 test at screening
* Hepatitis B Surface antigen negative
* Hepatitis C antibody negative, or if reactive, Hepatitis C RNA undetectable in plasma
* Volunteers born female of reproductive potential, sexually active with a male sex partner must agree to use one effective method of contraception from the time of signing the consent to completion of the study and agree to pregnancy testing as per the schedule of events.
* Study participants born female with reproductive potential are defined as pre-menopausal volunteers born female who have not had a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy). Volunteers born female are considered menopausal if they have not had a menses for at least 12 months and have an follicle stimulating hormone (FSH) of greater than 40 IU/L or if FSH testing is not available, they have had amenorrhea for 24 consecutive months.

Inclusion Criteria for HIV-1-Infected Viremic Subjects: Arm 3

* Aged >18 and <60 years at the time of screening
* Ability and willingness to provide written informed consent
* Willingness to comply with protocol schedule
* Willingness to undergo HIV-1 testing
* Reactive 4th generation point of care HIV-1 test at screening
* Plasma HIV-1 RNA levels > 2,000 copies/mL and < 100,000 copies/mL in subjects who are either:

  * ART-naïve
  * ART-experienced and in consultation with their primary provider have discontinued therapy for at least 8 weeks
  * ART-experienced, clinically stable and without changes to their ART regimen for at least 8 weeks
* Current CD4+ T cell count > 350 cells/mm3 and a nadir CD4+ T cell count > 250 cells/mm3
* Agrees not to begin or change antiretroviral therapy for 6 weeks after 10E8.4/iMab infusion despite a clear explanation of current Department of Health and Human Services (DHHS) guidelines
* Hepatitis B Surface antigen negative
* Hepatitis C antibody negative or if reactive Hepatitis C RNA undetectable in plasma
* Volunteers born female of reproductive potential, sexually active with a male sex partner agree to use one effective method of contraception from the time of signing the consent to completion of the study and agree to pregnancy testing as per the schedule of events.
* Study participants born female with reproductive potential are defined as pre-menopausal volunteers born female who have not had a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy). Volunteers born female are considered menopausal if they have not had a menses for at least 12 months and have an FSH of greater than 40 IU/L or if FSH testing is not available, they have had amenorrhea for 24 consecutive months.

Exclusion Criteria for HIV uninfected volunteers: Arms 1, 2 and 4:

* Confirmed HIV-1 infection
* At high risk of HIV-1 infection as defined by:

  * Unprotected intercourse with a casual or HIV-infected partner over the past 12 months
  * In a serodisconcordant relationship with an HIV-1 infected partner
  * A diagnosed new sexually transmitted infection within the past 12 months
  * Exchange of money or drugs for sex in the last 12 months
  * More than 2 sexual partners, defined as insertive or receptive vaginal or anal intercourse, within the past 6 months
* Weight above 100 kg at screening. Note that subjects above 80 kg may not be randomized into the SC dosing group in Arm 4.
* Any acute or chronic medical condition that in the opinion of the investigator would preclude participation
* Immunodeficiency or chronic autoimmune disease
* Intravenous drug use
* Excessive use of alcohol or recreational drugs that in the opinion of the investigator would preclude participation.
* Decompensated psychiatric illness
* Need for chronic immunotherapy including systemic corticosteroids, other monoclonal antibody therapy, or immunosuppressive drugs
* If born female, pregnant, lactating or planning on becoming pregnant over the study period
* Any of the following laboratory parameters:

  * Hemoglobin <10.0 g/dL
  * Absolute neutrophil count <1,000/mm3
  * Absolute lymphocyte count <500/mm3
  * Platelet count <100,000/mm3
  * Prothrombin time (PT) >1.25xULN
  * Partial thromboplastin time (PTT) >1.66xULN
  * Creatinine >1.25x Upper limit of normal (ULN)
  * Aminotransferase (AST) >1.5X ULN
  * Alanine Aminotransferase (ALT) >1.5X ULN
  * Glucose (non-fasting) >160mg/dL
  * Proteinuria: 2+ or greater
  * Hematuria: >10 RBC per high power field
  * Serum calcium < 8.5 mg/dL or >10.2 mg/dL
  * Serum parathyroid hormone (PTH) levels <10 pg/mL or >65 pg/mL
* Any vaccine administration within 14 days of study entry
* Experimental HIV-1 vaccine in past (active arm of an HIV-1 vaccine trial if applicable)
* Previous receipt of an experimental mAb to HIV-1 in a research study
* History of severe allergic reactions to drugs, vaccines, or drug infusion
* Participation in another investigational clinical trial within the past 12 weeks or anticipated during the course of the current study

Exclusion Criteria for HIV-1-Infected Viremic Subjects: Arm 3

* Any acute or chronic medical condition that in the opinion of the investigator would preclude participation
* A history of virologic failure of two or more combination antiretroviral treatment regimens. A regimen switch due solely to intolerance and not virologic failure does not qualify as a failed regimen.
* Weight above 100 kg at the time of screening.
* Intravenous drug use
* Excessive use of alcohol or recreational drugs that in the opinion of the investigator would preclude participation
* Decompensated psychiatric illness
* Need for chronic immunotherapy including systemic corticosteroids, other monoclonal antibody therapy, or immunosuppressive drugs
* If born female, pregnant, lactating or planning on becoming pregnant over the study period
* Any of the following laboratory parameters

  * Hemoglobin <10.0 g/dL
  * Absolute neutrophil count <1,000/mm3
  * Absolute lymphocyte count <500/mm3
  * Platelet count <100,000/mm3
  * PT >1.25xULN
  * PTT >1.66xULN
  * Creatinine >1.25x Upper limit of normal (ULN)
  * AST >1.5X ULN
  * ALT >1.5X ULN
  * Glucose (non-fasting) >160mg/dL
  * Proteinuria: 2+ or greater
  * Hematuria: >10 RBC per high power field
  * Serum calcium < 8.5 mg/dL and >10.2 mg/dL
  * Serum PTH level <10 pg/mL or >65 pg/mL
* Any vaccine administration within 14 days of study entry
* Experimental HIV-1 vaccine in past (active arm of an HIV-1 vaccine trial if applicable)
* Participation in a research study of a neutralizing monoclonal antibody (mAb) to HIV-1
* History of severe allergic reactions to drugs, vaccines, or drug infusion
* Participation in another investigational clinical trial within the past 12 weeks or anticipated during the course of the current study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Safety of the highest single intravenous dose of 10E8.4/iMab in HIV uninfected individuals. Safety of a single dose of intravenous dose of 10E8.4/iMab in HIV uninfected individuals | 24 weeks
  Percentage of subjects experiencing a dose limiting toxicity defined as a Grade 3 or 4 adverse events as per the toxicity grading scale for healthy volunteers enrolled in preventative vaccine trials
Safety of the highest single intravenous dose of 10E8.4/iMab in HIV infected individuals Safety of a single dose of intravenous dose of 10E8.4/iMab in HIV uninfected individuals | 24 weeks
  Percentage of subjects experiencing a dose limiting toxicity defined as a Grade 3 or more adverse event as per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events v 2.1
Injection site reactions associated with a single subcutaneous injection of 10 E8.4/iMab in HIV uninfected individuals | 24 weeks
  Percentage of injections associated with a Grade 2 or greater injection site reaction as per the toxicity grading scale for healthy volunteers enrolled in preventative vaccine trials
Systemic infusion reaction associated with the intravenous administration of any dose of 10E8.4/iMab | 24 weeks
  Percentage of subjects receiving intravenous 10E8.4/iMab as per CTCAE version 5.0.

SECONDARY OUTCOMES:
Antiviral activity of the highest single dose of 10E8.4/iMab given intravenously to viremic HIV infected individuals | 7 days
  changes in log HIV-1 RNA levels from baseline
Antiviral activity of the highest single dose of 10E8.4/iMab given intravenously to viremic HIV infected individuals | 14 days
  changes in log HIV-1 RNA levels from baseline
Antiviral activity of the highest single dose of 10E8.4/iMab given intravenously to viremic HIV infected individuals | 28 days
  changes in log HIV-1 RNA levels from baseline
Serum levels 10E8.4/iMab after the highest single dose of 10E8.4/iMab given intravenously to HIV infected and uninfected individuals | 7 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Serum levels of 10E8.4/iMab after the highest single dose of 10E8.4/iMab given intravenously to HIV infected and uninfected individuals | 14 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Serum levels of 10E8.4/iMab after the highest single dose of 10E8.4/iMab given intravenously to HIV infected and uninfected individuals. | 28 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Serum levels of 10E8.4/iMab after the highest single dose of 10E8.4/iMab given intravenously to HIV infected and uninfected individuals. | 56 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Serum levels of 10E8.4/iMab after the highest single dose of 10E8..4/iMab given subcutaneously to HIV uninfected individuals | 7 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Serum levels of 10E8.4/iMab after the highest single dose of 10E8..4/iMab given subcutaneously to HIV uninfected individuals | 14 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Serum levels of 10E8.4/iMab after the highest single dose of 10E8..4/iMab given subcutaneously to HIV uninfected individuals | 28 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Serum levels of 10E8.4/iMab after the highest single dose of 10E8..4/iMab given subcutaneously to HIV uninfected individuals | 56 days
  levels of 10E8.4/iMab expressed in ng/mL serum
Percentage of subjects developing antibodies to 10E8.4/iMab after any single intravenous or subcutaneous dose of 10E8.4/iMab | 84 days
  Percent of study participants

CONTACTS AND LOCATIONS:
Overall Officials: David D. Ho, MD, Principal Investigator — ADARC at CUIMC
Locations (2):
- United States (2):
  - Orlando Immunology Center, Orlando, Florida
  - Columbia University Research Unit, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hraber P, Seaman MS, Bailer RT, Mascola JR, Montefiori DC, Korber BT. Prevalence of broadly neutralizing antibody responses during chronic HIV-1 infection. AIDS. 2014 Jan 14;28(2):163-9. doi: 10.1097/QAD.0000000000000106. PMID 24361678
- [Background] Haynes BF, Gilbert PB, McElrath MJ, Zolla-Pazner S, Tomaras GD, Alam SM, Evans DT, Montefiori DC, Karnasuta C, Sutthent R, Liao HX, DeVico AL, Lewis GK, Williams C, Pinter A, Fong Y, Janes H, DeCamp A, Huang Y, Rao M, Billings E, Karasavvas N, Robb ML, Ngauy V, de Souza MS, Paris R, Ferrari G, Bailer RT, Soderberg KA, Andrews C, Berman PW, Frahm N, De Rosa SC, Alpert MD, Yates NL, Shen X, Koup RA, Pitisuttithum P, Kaewkungwal J, Nitayaphan S, Rerks-Ngarm S, Michael NL, Kim JH. Immune-correlates analysis of an HIV-1 vaccine efficacy trial. N Engl J Med. 2012 Apr 5;366(14):1275-86. doi: 10.1056/NEJMoa1113425. PMID 22475592